CLINICAL TRIAL: NCT05559541
Title: A Multicenter, Open-Label, Phase Ib/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of AK119 Combined With AK104 in Patients With Advanced Solid Tumors
Brief Title: Study of AK119 Combined With AK104 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development strategy adjustment
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK119-104
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK119+AK104 (Experimental): AK119 and AK104 IV every 2 or every 3 weeks.
  Interventions: Drug: AK119; Drug: AK104

INTERVENTIONS:
Drug: AK119 — AK119 is an anti-CD73 monoclonal antibody.
Drug: AK104 — AK104 is an anti-PD-1 and CTLA-4 bispecific antibody.

SUMMARY:
This is a Phase Ib/II Study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of AK119 combined with AK104 in tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign the written informed consent form (ICF) voluntarily.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status: 0 to1.
4. Life expectancy ≥12 weeks.
5. Subjects must have histologically or cytologically confirmed advanced solid tumor that is refractory or relapsed to the current standard therapies, or for which no effective standard therapy is available.
6. Subjects must have evaluable lesions according to RECIST v1.1.
7. Subjects must have adequate organ function.
8. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use effective barrier methods of contraception during the study and for 120 days after last dose of study drug.

Exclusion Criteria:

1. Prior malignancy active within the previous 3 years except for the locally curable cancers that have been apparently cured.
2. Being involved in another clinical study, except for observational clinical studies or follow-up period of interventional studies.
3. Have exposed to other products targeting T cell costimulation or immune checkpoint pathway excepts for PD-1/PD-L1 inhibitor.
4. Anticancer therapy (e.g., chemotherapy, radiotherapy, etc.) within 4 weeks prior to the first dose of investigational product; Anticancer small-molecule targeted agent (e.g., tyrosine kinase inhibitor) within 2 weeks prior to the first dose of investigational product.
5. Subjects with spinal cord compression or active brain metastases, except for subjects with untreated and asymptomatic brain metastases or with stable brain metastases after treatment.
6. Subjects with pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
7. Subjects whose imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the study.
8. Toxicities of prior anticancer therapy have not resolved to ≤ Grade 1 (NCI-CTCAE version 5.0).
9. Patients with clinically significant cardio-cerebrovascular or venous thromboembolic disease.
10. Active autoimmune diseases or history of autoimmune diseases that may relapse.
11. History of interstitial lung disease or noninfectious pneumonitis.
12. Major surgery or trauma within 4 weeks prior to first dose of investigational product. Unhealed wound, ulcer or fracture within 4 weeks prior to first dose of investigational product.
13. Any condition that required systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of investigational product.
14. Receipt of live attenuated vaccines within 4 weeks prior to the first dose of investigational product.
15. Previous history of severe hypersensitivity reactions to other monoclonal antibodies.
16. Patients are pregnant or breastfeeding, or plan to breastfeed during the study.
17. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation.
18. Any other conditions that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | During the first 3 or 4 weeks
  DLTs will be assessed during the first 3 or 4 weeks of treatment. DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT observation period.
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug.
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with CR or PR (based on RECIST Version 1.1).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST Version 1.1).
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST Version 1.1).
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to 2 years
  Time to response (TTR) is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR (based on RECIST Version 1.1).
Overall survival (OS) | Up to 2 years
  OS defined as the time from the first dose to death from any cause.
PK parameters | From first dose of study drug through last dose
  The PK parameters include serum concentrations of AK119 and AK104 at different timepoints after study drug administration.
Immunogenicity assessment | From first dose of study drug through 30 days after last dose
  The immunogenicity of AK119 and AK104 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, PhD, Principal Investigator — Tianjin Medical University Cancer Insitute & Hospital
Locations (1):
- Tianjin Medical University Cancer Insitute & Hospital, Tianjin, Tianjin Municipality, China